CLINICAL TRIAL: NCT04623398
Title: Effect of Lithium in Patients With Autism Spectrum Disorder and Phelan-McDermid Syndrome (SHANK3 Haploinsufficiency): Pilot Study.
Brief Title: Effect of Lithium in Patients With Autism Spectrum Disorder and Phelan-McDermid Syndrome (SHANK3 Haploinsufficiency)
Acronym: Lisphem
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160914J
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; Lithium
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium (Experimental): Li+ is an FDA (NDA: 016834) and ANSM (AMM 3400931376339) approved drug. There are two lithium salts that are marketed in France, Teralithe LI (cp 250mg) and Teralithe LP (cp 400mg).
  The experimental drugs in this study will be lithium carbonate capsules dosed at 62.5mg, 125mg and 250mg prepared as hospital preparations for clinical trials.
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator): Capsules containing lactose monohydrate in all points resembling the capsules of active ingredients.
  Capsules of pla62.5 mg, pla125 mg and pla250 mg (pla=placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — The experimental drugs in this study will be lithium carbonate capsules dosed at 62.5mg, 125mg and 250mg prepared as hospital preparations for clinical trials.
  Arms: Lithium
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
There is currently no treatment for the body symptoms of Autism Spectrum Disorders (ASD). However, basic research suggests that some forms of ASD may be alleviated, even in the adult stage. The genes involved in ASDs particularly impact synaptic homeostasis. Specific clinical trials in patients with synaptic mutations need to be carried out. In this spirit, patients with deleterious mutations in SHANK3 represent a paradigm. The induced pluripotent stem cells (iPSc) carrying SHANK3 mutations and derived in neurons, can be used for high-throughput screening of pharmacological substances and allow the identification of compounds that can restore the expression level of SHANK3. The objective of this proposed project is to test one of the compounds identified by research on these iPSc as a novel treatment for social communication deficit in patients with deleterious mutations in SHANK3. Its effect on the symptoms of the social deficit could represent a new perspective for other forms of idiopathic autism.

DETAILED DESCRIPTION:
Phase IIa intervention study, pilot, prospective, multicenter, randomized in 2 parallel arms, Li+ versus placebo, double-blind. The main objective of the study is to evaluate the effect of Li+ at 12 weeks, compared to placebo, on the social communication deficit in patients with Phelan-McDermid Syndrome (SHANK3 haploinsufficiency).

The Secondary Objectives are :

* To evaluate the effect of Li+ at 12 weeks on all cardinal and main symptoms in patients suffering from Phelan-McDemid Syndrome (PMS).
* Evaluate the tolerance of Li + for 12 weeks in children suffering from PMS.
* Demonstrate the feasibility of a phase III, randomized controlled trial.
* Evaluate the residual effect of treatment at 16 to 18 weeks after stopping treatment)
* Evaluate the parents' feelings at the end of the study regarding the child's behavior and the impact on their daily lives

The treatment of the study is lithium carbonate: Li+ carbonate capsules are prepared from the raw material for pharmaceutical use .

Inclusion will be ensured by the clinical genetics centers. Psychiatric evaluation will be carried out by the investigative child psychiatry service.

Patients will be followed up by 2 referring physicians:

* a child psychiatrist, blind of the treatment arm, who will carry out the evaluations of the judgement criteria;
* a physician from the clinical investigation center, the only one informed of the attribution arm, who will ensure the adaptation of the LI dosage; an adaptation of the dummy dosage will be proposed to the patients on placebo to maintain the blind in this group as well. A lithiaemia will be performed every 4 days (+/- 1 day) until the target lithiaemia of 0.4-0.6 meq/L is reached with progressive increment of the lithium dose administered. The target blood lithium level must be reached within 20 days

As the evaluation is based on hetero-evaluation (by the parents), a placebo treatment remains necessary in the control arm.

Pharmaceutical preparations will be carried out for this pilot study: unit blister packaging of the active ingredient and the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years of age
* Minimum weight of 20 kg for children aged 7 years old
* Patient with haplo deficiency SHANK3, i.e. carrier of a SHANK3 deletion (CNV) or a de novo truncating mutation in SHANK3 (Phelan McDermid syndrome);
* Total Social Responsiveness Scale - T score (SRS) of at least 66
* Patients of childbearing age who are sexually active must agree to use a highly effective form of contraception (estrogen-progestin or progestin-only contraception, or an intrauterine device, or contraceptive abstinence).
* Affiliation to a social security system
* Signature of the consent by the holders of parental authority
* Non-participation in another clinical trial
* Diagnosis of Autism Spectrum Disorders (DSM-5 criteria) confirmed by Autism Diagnostic Interview-Revised (ADI-R) and Autism Diagnostic Observation Scale (ADOS-II)
* IQ Assessment
* Beta-HCG negative

Exclusion Criteria:

* Hepatic or renal insufficiency (disturbed liver function tests, abnormal creatinine clearance);
* Unbalanced thyroid or diabetic pathology;
* Cardiac pathology: Brugada syndrome or family history of Brugada syndrome, heart failure;
* Addison's disease;
* Unstable epileptic disease.
* Patient with concomitant diseases judged for which the experimental treatment with Li + could compromise tolerance ;
* History of allergy to Li+;
* Allergy to lactose, lactose being the sole diluent and excipient of the prepared form.
* Initiation of co-occurring cognitive-behavioural therapy that is specifically focused on autistic symptoms within 6 weeks prior to inclusion;
* Any introduction of psychotropic drugs within 2 weeks prior to trial, including neuroleptics, monoamine oxidase inhibitors, stimulants, antidepressants. For neuroleptic drugs and Fluoxetine, this delay should be 4 weeks prior to the trial;
* Serious behavioural problems or refusal to take medication that does not allow for compliance;
* Inability to perform blood tests to check lithemia when the patient is included.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Score social responsiveness scale | 12 weeks
  Severity of Autistic Symptoms - Social Responsiveness Scale - Total score at 12 weeks.

SECONDARY OUTCOMES:
Score social responsiveness scale | Baseline (At randomization) , 4 weeks, 8 weeks, and 16 to 18 weeks after stopping the treatment
  Severity of Autistic Symptoms - Social Responsiveness Scale. Evaluate the effect of the treatment on the severity of autistic symptoms.
  Exploring the improvement of cardinal autistic symptoms (particularly social communication) during the therapeutic trial.
score of autism diagnosis observation scale | Baseline (At randomization) and 12 weeks
  Autism Diagnosis Observation Calibrated Severity Score. Evaluate the effect of the treatment on the improvement of cardinal autistic symptoms (particularly social communication) during the therapeutic trial.
Score of attention deficit hyperactivity disorder | Baseline (At randomization) 4 weeks, 8 weeks, 12 weeks, and 16 to 18 weeks after stopping the treatment
  assessment of hyperactivity. Evaluate the effect of the treatment on the improvement of cardinal autistic symptoms (particularly social communication) during the therapeutic trial.
score of child's sleep disorder rating scale | Baseline (At randomization) , 4 weeks, 8 weeks, 12 weeks and 16 to 18 weeks after stopping the treatment
  Evaluate the effect of the treatment on Child's Sleep Disorder
Score of Dunn Sensory Profile | 4 weeks, 8 weeks, 12 weeks and 16 to 18 weeks after stopping the treatment
  Evaluate the effect of the treatment on the improvement of cardinal autistic symptoms (particularly social communication) during the therapeutic trial.
Score of Aberrant Behavior checklist scale | Baseline (At randomization), 4 weeks, 8 weeks and 12 weeks
  Aberrant Behavior Checklist Scale - Social Withdrawal Subscale. Exploring aberrant, stereotyped, repetitive and obsessive behaviours (sub-scores and total score) and co-morbidities
score of global functioning | Baseline (At randomization), 4 weeks, 8 weeks, 12 weeks and 16 to 18 weeks after stopping the treatment
  Clinical Global Improvement - Improvement and Severity Scores. Evaluate the effect of the treatment on the global functioning of patients and the impact on their environment
Score of Vineland Adaptive Behavior Composite | Baseline (At randomization) and12 weeks
  Evaluate the effect of the treatment on the global functioning of patients and the impact on their environment
Score of surrounding constraints | Baseline (At randomization), 4 weeks, 8 weeks, 12 weeks and 16 to 18 weeks after stopping the treatment
  Surrounding Constraints - Caregiver Strain Index. Evaluate the effect of the treatment on the global functioning of patients and the impact on their environment
score of Columbia Suicide Severity Rating Scale | Baseline (At randomization)and 12 weeks
  Monitoring suicide risk and suicidal risk via the Columbia Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Delorme Richard, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France